CLINICAL TRIAL: NCT02441348
Title: Efficacy of Conversation Training Therapy (CTT)
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Jacqueline Gartner-Schmidt, Professor, University of Pittsburgh
Other Study IDs: PRO15030497
Record Dates: First submitted 2015-05-06; First posted 2015-05-12 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Voice Disorders
Keywords: Voice Therapy; Muscle Tension Dysphonia; Lesions
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CTT group: CTT will be initiated in a prospective fashion to study population
  Interventions: Behavioral: Conversation Training Therapy

INTERVENTIONS:
Behavioral: Conversation Training Therapy — Conversational speech as the primary focus of voice therapy in individuals with muscle tension dysphonia or vocal fold lesions.

SUMMARY:
Voice therapy is the standard-of-care for many of the nearly 140 million people in the United States who suffer from voice disorders,1 yet patients claim that current therapies are ineffective at meeting their voice needs.2 Published data by our research team indicate that patients think that transfer of target voice techniques to every day voice use (i.e. conversation) is the most difficult aspect of therapy,2 and that training techniques in conversation is the most useful aspect of voice therapy.2 Unfortunately, traditional voice therapy programs spend little, if any, time training voice techniques in conversation.3 This lack of functional specificity in voice therapy may contribute to the estimated 65% attrition rate.4 Even after some form of treatment, patients are still struggling with daily conversational voice use, and voice disorders continue to cause serious disability, stress and depression, which negatively affects social functioning and job performance.5 A new voice therapy program, Conversation Training Therapy (CTT), based on published patient reports on dissatisfaction with traditional therapy, was developed by the Investigators. It was honed with recommendations from expert clinical voice-specialized speech-language pathologists, and successfully piloted in a small case series of patients with voice problems. The investigators objective in this application is to test CTT in the rehabilitation of patients with voice disorders. The investigators hypothesize that, as demonstrated in the investigators preliminary case studies, these methods will result in early treatment success, and reduce the time required to reach therapeutic goals, thereby reducing costs associated with voice treatment.

DETAILED DESCRIPTION:
Two common voice disorders, vocal fold lesions (lesions) and muscle tension dysphonia (MTD) constitute over 60% of voice clinic caseloads. Over 80% of patients with lesions and nearly 100% of those with MTD are treated exclusively with voice therapy.7,8 Traditional, bottom-up hierarchical, non-conversation based voice therapy is the established standard of care used most widely by speech-language pathologists (SLP) in clinical practice.e.g.3,9,10 However, the investigators group's published research indicated a clear need to target conversational voice use in treatment.2 Currently, no treatment program exists with a focus on voice use in conversation. Most voice therapy techniques are based in hierarchical, programmatic approaches aimed at manipulating phonatory physiology for voice improvement. These hierarchies necessitate that the final step in therapy is generalization of the target voice techniques to spontaneous, conversational speech.3 Three major problems exist with this approach to voice therapy, which the current proposal aims to address.

First, A hierarchical non-conversational approach to therapy builds treatment from unvoiced breathing to single sounds and rote phrases to connected speech to spontaneous every day conversation last, if at all, and patients are often discharged from therapy unable to generalize therapy techniques to conversation. Second, the use of a hierarchical, bottom-up approach necessitates a protracted time in treatment. Third, attrition rates for behavioral voice therapy are estimated between 16-65%,4,17 and voice problem relapse rates are between 51-68%.

ELIGIBILITY:
Inclusion Criteria:

* males and females
* age 18-60 years old
* diagnosed by a multi-disciplinary team consisting of laryngologist and speech-language pathologist with muscle tension dysphonia (MTD) or vocal fold lesions deemed amenable to voice therapy (i.e. not surgical candidates) using a standardized stimulability test developed by the research team (in revision for publication)

Exclusion Criteria:

* age 61 or greater
* under 18 years of age

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Individuals diagnosed with either muscle tension dysphonia (MTD) or vocal fold lesion who are candidates for voice therapy.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09-27 (Actual)

PRIMARY OUTCOMES:
Change in the Voice Handicap Index-10 (VHI-10) | Baseline through completion of therapy; approximately 6-8 months

CONTACTS AND LOCATIONS:
Overall Officials: Amanda I Gillespie, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided